CLINICAL TRIAL: NCT06023147
Title: A Real-world Study of the Short-term Efficacy and Safety of Elaboration Transcatheter Arterial Chemoembolization (E-TACE) in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: A Real-world Study of the Short-term Efficacy and Safety of E-TACE in Patients With Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, Associate Professor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-0737-002
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: E-TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-TACE (Experimental): Procedure: The 100μm drug-loaded microspheres were loaded with 40mg-80mg anthracyclines at one milliliter/two milliliter (1mL/2mL), and then combined with non-isoionic contrast agents to embolize the tumor supplying arteries, and then 250μm or 400μm drug-loaded microspheres were loaded with 1mL/2mL chemotherapy drugs to embolize the tumor supplying arteries at different grades and diameters.
  Interventions: Procedure: E-TACE

INTERVENTIONS:
Procedure: E-TACE — The 100μm drug-loaded microspheres were loaded with 40mg-80mg anthracyclines at 1mL/2mL, and then combined with non-isoionic contrast agents to embolize the tumor supplying arteries, and then 250μm or 400μm drug-loaded microspheres were loaded with 1mL/2mL chemotherapy drugs to embolize the tumor supplying arteries at different grades and diameters.

SUMMARY:
This is a real world study to determine the short-term efficacy and safety of Elaboration transcatheter arterial chemoembolization (E-TACE) for hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Primary liver cancer is the fourth common malignant tumor and the second cause of death in China, which seriously threatens the life and health of Chinese people. Hepatocellular carcinoma accounts for 75% to 85% of primary liver cancer and is considered the leading cause of death in patients with cirrhosis, and its incidence is expected to continue to increase.

At present, the main treatment methods of liver cancer are surgical resection, liver transplantation, interventional therapy, etc., HCC patients are often advanced in initial diagnosis, coupled with cirrhosis, liver function intolerance and other factors, only about 15% of patients can receive surgical resection. Transcatheter arterial chemoembolization (TACE) has been applied in hepatocellular carcinoma for more than 40 years. TACE treatment can be divided into conventional TACE and Drug-eluting beads-transarterial chemoembolization (DEB-TACE) according to different embolic agents. DEB-TACE refers to the embolization therapy based on drug-eluting microspheres loaded with chemotherapy drugs, which can embolize the blood supplying artery of liver cancer to cause tumor ischemia and necrosis. At the same time, as a carrier of chemotherapy drugs, DEB-TACE has the advantage of continuously and steadily releasing drugs, so that the local tumor can reach a higher required concentration. Elaboration transcatheter arterial chemoembolization (E-TACE) is the elaboration transcatheter arterial branch selection of the tumor and the refined embolization is carried out by using uniform drug-loaded microsphere.

Although there have been a large number of randomized controlled studies on TACE treatment of HCC, due to the clear inclusion or exclusion criteria of randomized controlled studies. The results of the studies are different from the real diagnosis and treatment environment due to the limitations of treatment programs. This difference is called the efficacy effectiveness gap (EEG). In addition, the 2022 edition of China Liver Cancer Standard Diagnosis and Treatment Quality Control Indicators and 2022 edition of Primary Liver Cancer Diagnosis and Treatment Guidelines point out that TACE treatment for liver cancer needs to be standardized and refined, to reduce the heterogeneity of tumors leading to differences in TACE efficacy, and ultimately improve the survival rate and survival habits of liver cancer patients. There are currently no real-world studies on the efficacy and safety of E-TACE in the treatment of hepatocellular carcinoma. Therefore, this study intends to conduct a real-world study to evaluate the short-term efficacy and safety of E-TACE in the treatment of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Gender and age are not limited;
2. HCC patients who strictly meet the clinical diagnostic criteria of the Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2022 edition) or who have been confirmed by histopathology or cytology;
3. Patients who have at least one tumor supply artery available for superselection, and who are assessed by investigators or multi-disciplinary treatment (MDT) to require E-TACE therapy;
4. Patients sign informed consent and have good compliance.

Exclusion Criteria:

1.Patients judged by the investigators to be unsuitable for inclusion in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1, 3, 6,12 months after the first E-TACE treatment, up to death or 12 months
  Proportion of patients with reduction in stable in tumor burden of a predefined amount

SECONDARY OUTCOMES:
6/12 months progression-free survival (PFS) rate | 6/12 months
  Rate of progression free survival in 6/12 months
6/12 months overall survival (OS) rate | 6/12 months
  Rate of over survival rate in 6/12 months
Disease control rate (DCR) | 1, 3, 6,12 months after the first E-TACE treatment, up to death or 12 months
  Proportion of patients with reduction or keeping in stable in tumor burden of a predefined amount

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Duan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (27):
- China (27):
  - Huai He Hospital of Henan University, Kaifeng, Henan
  - Luo He Central Hospital, Luohe, Henan
  - WuYang People's Hospital, Luohe, Henan
  - Luo Yang Central Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Deng zhou People's Hospital, Nanyang, Henan
  - First People's Hospital of Ping Dingshan, Pingdingshan, Henan
  - General Hospital of Pingmei Shenma Group, Pingdingshan, Henan
  - Lushan Xian People's Hospital, Pingdingshan, Henan
  - Second People's Hospital of Ping Dingshan, Pingdingshan, Henan
  - The 989 Hospital of the Chinese People's Liberation Army Joint Logistic Support Force, Pingdingshan, Henan
  - Puyang People's Hospital, Puyang, Henan
  - San Menxia Central Hospital, Sanmenxia, Henan
  - Yellow River San Menxia Hospital, Sanmenxia, Henan
  - Central Hospital of Yongcheng, Shangqiu, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - Shangqiu Municipal Hospital, Shangqiu, Henan
  - The People's Hospital of Yongcheng, Shangqiu, Henan
  - Tumor Hospital of Xinyang, Xinyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Sixth Peoples Hospital of Zhengzhou, Zhengzhou, Henan
  - The Third Peoples Hospital of Zhengzhou, Zhengzhou, Henan
  - First People's Hospital of Zhoukou, Zhoukou, Henan
  - Xihua Xian People's Hospital, Zhoukou, Henan
  - Zhou Kou Central Hospital, Zhoukou, Henan
  - Zhou Kou Hospital of TCM, Zhoukou, Henan